CLINICAL TRIAL: NCT04008082
Title: Specific Use Results Survey of LENVIMA 4 mg Capsules -Observational Study of Overall Survival in Patients With Unresectable Hepatocellular Carcinoma (Study LEN03T)
Brief Title: A Study of Overall Survival in Participants With Unresectable Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7080-M081-510; LEN03T (Other: EISAI)
Record Dates: First submitted 2019-05-13; First posted 2019-07-05 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-06

CONDITIONS: Carcinoma, Hepatocellular; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms
Keywords: Hepatocellular Carcinoma; Lenvatinib Mesilate; Lenvima; LEN03T
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lenvatinib: Lenvatinib capsules 12 milligram (mg) for participants with body weight greater than or equal to (>=) 60 kilograms (kg) or 8 mg for participants with body weight less than (<) 60 kg, orally, once daily as per routine clinical practice.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsule.
  Other Names: Lenvima; E7080

SUMMARY:
The primary purpose of this study to continue follow-up of participants enrolled in the study E7080-M081-504 (NCT03663114) of lenvima capsules and to evaluate the overall survival of participants with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

- All participants enrolled in the study E7080-M081-504 with informed consent to participate in this study.

Exclusion Criteria:

* Participants who do not have unresectable hepatocellular carcinoma
* Participants who have not given informed consent or have withdrawn consent to participation
* Participants with a history of hypersensitivity to any ingredient of lenvima
* Pregnant or possibly pregnant women
* Participants previously treated with lenvima (excluding those previously enrolled in the Study E7080-M081-504 [NCT03663114] at another clinical site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with unresectable hepatocellular carcinoma will be observed for specific use results survey of lenvima 4 mg capsules.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of study drug administration until date of death from any cause (approximately 2.8 years)
  OS is calculated as the period from the day of starting administration to the day of death from any cause.
Presence or absence of factors with a possible influence on OS | From date of study drug administration until date of death from any cause (approximately 2.8 years)
  Factor analysis is performed according to the category of participant background (aetiology of chronic liver disease, baseline alpha-fetoprotein concentration etc), lenvima administration status and treatment situation before and after administration of lenvima, and factors affecting OS are examined. Appropriate statistical methods (Cox regression analysis, etc.) will be used to examine the relationship of OS with various factors in order to identify the factors affecting survival.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Eisai Trial Site #1, Osaka
  - Eisai Trial Site #2, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Furuse J, Izumi N, Motomura K, Inaba Y, Katamura Y, Kondo Y, Yabushita K, Matsuoka T, Motoyoshi K, Kudo M. Long-Term Survival of Patients with Unresectable Hepatocellular Carcinoma Treated with Lenvatinib in Real-World Clinical Practice. Cancers (Basel). 2025 Feb 1;17(3):479. doi: 10.3390/cancers17030479. PMID 39941845